CLINICAL TRIAL: NCT02989480
Title: PET-detected Myocardial Inflammation is a Characteristic of Cardiac Sarcoid But Not of ARVC - a Feasibility Study
Brief Title: PET-detected Myocardial Inflammation is a Characteristic of Cardiac Sarcoid But Not of ARVC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 3/072/14
Record Dates: First submitted 2016-01-20; First posted 2016-12-12 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Sarcoidosis; Arrhythmogenic Right Ventricular Cardiomyopathy
Keywords: Cardiomyopathy
MeSH Terms: conditions — Sarcoidosis; Arrhythmogenic Right Ventricular Dysplasia; Cardiomyopathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — ACE inhibitors and CRP will be measured.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sarcoidosis: Patients with cardiac sarcoidosis diagnosed according to the Japanese Ministry of Health and Welfare criteria will be included. All patients will have histologically proven sarcoidosis (cardiac biopsy not mandatory) and no other potential cardiac disease. They will have no family history of cardiomyopathy.
  Interventions: Radiation: PET CT; Other: Cardiac MRI
- Arrhythmogenic RV cardiomyopathy: Patients with ARVC diagnosed according to the Task Force criteria with in addition either a positive family history for the condition or harbour a known pathological mutation associated with it.
  Interventions: Radiation: PET CT; Other: Cardiac MRI

INTERVENTIONS:
Radiation: PET CT — PET CT scans
Other: Cardiac MRI — Cardiac MRI

SUMMARY:
Arrhythmogenic right ventricular cardiomyopathy (ARVC) is a rare condition in which the heart muscle cells especially of the main pumping chamber (the 'ventricle') is replaced by fat and scar tissue. Sarcoidosis is a condition that can affect many organs but when it affects the heart patches of inflammation can result in scarring, especially of the ventricles. Both conditions can cause dangerous heart rhythms and sudden death. Sarcoidosis can be treated with inflammation suppressing treatment (steroids), as well as pacemakers and implantable defibrillators which shock the heart back to normal rhythm. ARVC is usually treated with implantable defibrillators. The diagnosis of either condition can be difficult and indeed distinguishing the two can be extremely challenging. Increasingly nuclear scans (PET) are used to identify inflammation in the heart in patients suspected of having cardiac sarcoid. It is not known whether patients with ARVC have abnormal PET scans.

DETAILED DESCRIPTION:
Arrhythmogenic right ventricular cardiomyopathy (ARVC) is a rare inherited condition characterised pathologically by fibro-fatty replacement of myocytes usually (but not exclusively) within the right ventricle. The clinical consequences of this process are usually re-entrant ventricular arrhythmias which may be fatal and ARVC consequently is the third most common cause of sudden cardiac death in the young. Diagnosis involves imaging, electrocardiography, myocardial biopsy and genetic testing. Task Force criteria for the diagnosis have been established. Nevertheless the condition can be difficult to diagnose (or exclude), especially in less advanced disease, a common scenario in individuals with a family member suffering from the condition. To complicate the situation further, we and others have published recent reports suggesting that other infiltrative conditions within the heart especially sarcoidosis, may fulfil Task Force criteria, leading to a false positive diagnosis. This is a particular concern since the natural history and treatment options for these conditions are very different.

Sarcoidosis is a granulomatous disorder of unknown cause, predominantly affecting the lungs, reticuloendothelial systems and skin. Cardiac involvement at autopsy is found in up to 25% of affected individuals although clinical manifestations are only present in approximately 5%. Isolated cardiac sarcoidosis, without manifestations in other systems is rare. The non-caseating granulomas frequently infiltrate left ventricular & septal myocardium although right ventricular involvement also occurs. Granulomas and resulting scar formation can cause conduction disturbances, cardiac failure and ventricular arrhythmias. Sudden death is not uncommon. Myocardial biopsy confirms the diagnosis but because of the patchy nature of the granulomatous process, the test is only positive in 50% of the affected individuals. Other investigations used to help make or support the diagnosis include echocardiography, MRI, electrocardiography, PET, and corroborating evidence from high resolution CT chest and skin biopsy. However, imaging findings may lack specificity for a precise aetiology. Cardiac MRI identifies areas of myocardial scar or fibrosis, which is the final step in the disease process. Although patterns of fibrosis have been well described in ARVC and cardiac sarcoidosis, significant overlap exists between these two diseases with regard to the exact location of fibrosis: for example ARVC can affect either or both ventricles. Typically, although affecting predominantly the RV, in advanced stages there is also a well described pattern of mid-wall patchy fibrosis in the basal infero-lateral wall of the left ventricle and sometimes in the inter-ventricular septum. Conversely, sarcoidosis typically affects the LV, and when fibrosis is found, the location is in the septal or infero-lateral territories. In sarcoid, RV enlargement can occur either due to granulomatous involvement within the RV myocardium, or secondary to the pulmonary hypertension associated with lung involvement. Cases of sarcoidosis where the RV is involved may be more difficult to diagnose: The RV enlargement and reduction in function overlap significantly with the Task Force Criteria for the CMR diagnosis of ARVC, furthermore, the pattern of late gadolinium enhancement is not sufficiently specific to guide the diagnosis to either ARVC or Cardiac Sarcoid with RV involvement.

ELIGIBILITY:
Inclusion Criteria:

* Twenty patients from the age of 18-70 will be studied. We will include 10 patients with cardiac sarcoidosis diagnosed according to the Japanese Ministry of Health and Welfare criteria. All patients will have histologically proven sarcoidosis (cardiac biopsy not mandatory) and no other potential cardiac disease. They will have no family history of cardiomyopathy. We will also study 10 patients with ARVC diagnosed according to the Task Force criteria with in addition either a positive family history for the condition or harbour a known pathological mutation associated with it.

Exclusion Criteria:

* patients outside the age limit defined above and those who do not fulfil our inclusion criteria for either cardiac sarcoidosis or ARVC will be excluded.
* unwillingness to participate
* patients with any contraindication to MR scanning
* pregnant or breast feeding women
* diabetes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty patients from the age of 18-70 will be studied. We will include 10 patients with cardiac sarcoidosis diagnosed according to the Japanese Ministry of Health and Welfare criteria. All patients will have histologically proven sarcoidosis (cardiac biopsy not mandatory) and no other potential cardiac disease. They will have no family history of cardiomyopathy. We will also study 10 patients with ARVC diagnosed according to the Task Force criteria with in addition either a positive family history for the condition or harbour a known pathological mutation associated with it.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-08; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Myocardial inflammation or fibrosis by cardiac MRI and PET CT | Three hours
  Cardiac MRI and PET CT

CONTACTS AND LOCATIONS:
Overall Officials: Paul Broadhurst, Consultant, Principal Investigator — NHS Grampian
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, Aberdeenshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marcus FI, McKenna WJ, Sherrill D, Basso C, Bauce B, Bluemke DA, Calkins H, Corrado D, Cox MG, Daubert JP, Fontaine G, Gear K, Hauer R, Nava A, Picard MH, Protonotarios N, Saffitz JE, Sanborn DM, Steinberg JS, Tandri H, Thiene G, Towbin JA, Tsatsopoulou A, Wichter T, Zareba W. Diagnosis of arrhythmogenic right ventricular cardiomyopathy/dysplasia: proposed modification of the task force criteria. Circulation. 2010 Apr 6;121(13):1533-41. doi: 10.1161/CIRCULATIONAHA.108.840827. Epub 2010 Feb 19. PMID 20172911
- [Background] Dempsey OJ, Paterson EW, Kerr KM, Denison AR. Sarcoidosis. BMJ. 2009 Aug 28;339:b3206. doi: 10.1136/bmj.b3206. No abstract available. PMID 19717499
- [Background] Mohsen A, Panday M, Wetherold S, Jimenez A. Cardiac sarcoidosis mimicking arrhythmogenic right ventricular dysplasia with high defibrillation threshold requiring subcutaneous shocking coil implantation. Heart Lung Circ. 2012 Jan;21(1):46-9. doi: 10.1016/j.hlc.2011.08.013. Epub 2011 Oct 6. PMID 21982156
- [Background] Sen-Chowdhry S, Morgan RD, Chambers JC, McKenna WJ. Arrhythmogenic cardiomyopathy: etiology, diagnosis, and treatment. Annu Rev Med. 2010;61:233-53. doi: 10.1146/annurev.med.052208.130419. PMID 20059337
- [Background] Patel MR, Cawley PJ, Heitner JF, Klem I, Parker MA, Jaroudi WA, Meine TJ, White JB, Elliott MD, Kim HW, Judd RM, Kim RJ. Detection of myocardial damage in patients with sarcoidosis. Circulation. 2009 Nov 17;120(20):1969-77. doi: 10.1161/CIRCULATIONAHA.109.851352. Epub 2009 Nov 2. PMID 19884472
- [Background] Lobert P, Brown RK, Dvorak RA, Corbett JR, Kazerooni EA, Wong KK. Spectrum of physiological and pathological cardiac and pericardial uptake of FDG in oncology PET-CT. Clin Radiol. 2013 Jan;68(1):e59-71. doi: 10.1016/j.crad.2012.09.007. Epub 2012 Nov 22. PMID 23177651
- [Background] Campian ME, Verberne HJ, Hardziyenka M, de Groot EA, van Moerkerken AF, van Eck-Smit BL, Tan HL. Assessment of inflammation in patients with arrhythmogenic right ventricular cardiomyopathy/dysplasia. Eur J Nucl Med Mol Imaging. 2010 Nov;37(11):2079-85. doi: 10.1007/s00259-010-1525-y. Epub 2010 Jul 6. PMID 20603720
- [Background] Soejima K, Yada H. The work-up and management of patients with apparent or subclinical cardiac sarcoidosis: with emphasis on the associated heart rhythm abnormalities. J Cardiovasc Electrophysiol. 2009 May;20(5):578-83. doi: 10.1111/j.1540-8167.2008.01417.x. Epub 2009 Jan 9. PMID 19175448
- [Background] Williams G, Kolodny GM. Suppression of myocardial 18F-FDG uptake by preparing patients with a high-fat, low-carbohydrate diet. AJR Am J Roentgenol. 2008 Feb;190(2):W151-6. doi: 10.2214/AJR.07.2409. PMID 18212199
- [Background] Langah R, Spicer K, Gebregziabher M, Gordon L. Effectiveness of prolonged fasting 18f-FDG PET-CT in the detection of cardiac sarcoidosis. J Nucl Cardiol. 2009 Sep-Oct;16(5):801-10. doi: 10.1007/s12350-009-9110-0. Epub 2009 Jun 23. PMID 19548047